CLINICAL TRIAL: NCT04439825
Title: Randomized Controlled Single Blind Cross Over Trial Evaluating the Impact of Botox Treatment Into the Upper One Third of the Face an Area on Mood and Self -Appearance Satisfaction in a Post Covid Period.
Brief Title: Impact of Botox Treatment Into the Upper One Third of the Face an Area on Mood and Self -Appearance Satisfaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BTX-PST-COVID
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Mood
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botox (Active Comparator)
  Interventions: Drug: Botulinum Neurotoxin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Neurotoxin — glabella, forehead lines and/or lateral canthal lines
  Arms: Botox
Drug: Placebo — Saline solution (preservative free)
  Arms: Placebo

SUMMARY:
Botox treatment into the upper one third of the face (glabella, forehead lines and/or lateral canthal lines) to analyze mood and self -appearance satisfaction in a Post Covid period on non-naïve Botox patients

DETAILED DESCRIPTION:
A historical period that will never happen again provides us a unique opportunity to evaluate the impact Botox Cosmetic has on the mood and self appearance satisfaction after a societal crisis such as the COVID19 pandemic.

Many regular users of Botox Cosmetic will have exceeded their normal treatment interval and their glabellar wrinkles will likely have returned to baseline. Many will want to get treated as soon as stay at home orders are rescinded and clinics are permitted to open back up. It would not be surprising that these patients also are experiencing a decrease in their mood secondary to weeks of social isolating and distancing. Many can expect to have a rebound elevation in their happiness and overall mood following the modified return to normalcy.

Botox Cosmetic has been studied as a mood elevating drug by reducing the animation of a glabellar furrow via the facial feedback mechanism hypothesis. This has been shown in patients who are not diagnosed with a major depressive disorder. Following a natural disaster, does the administration of Botox Cosmetic, in patients who are frequent Botox Cosmetic users, synergistically amplify the elevation in mood beyond what would be achieved had they not had their Botox Cosmetic treatment. Perhaps regular Botox Cosmetic users have a secondary gain desire for Botox Cosmetic beyond wrinkle reduction but also as a mood elevator.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18-75
* Subjects will be non-naive Botox users with a glabellar wrinkle severity score of 2 or 3 who are at least 20 weeks from their last BOTOX Cosmetic treatment
* Subjects that understand the purpose and aspects of the study, freely sign the consent and complete the required treatment and follow up visits.

Exclusion Criteria:

* Males and females below the age of 18
* Subjects that received neuromodulator injections to the glabella region in the last 20 weeks
* Subjects who do not meet a 2-3 wrinkle severity score in the glabellar region
* Subjects who have received other invasive or semi invasive cosmetic forehead or glabellar treatments
* Subjects who have had a change in antidepressant or anti- anxiety medication in last 6 weeks
* Subjects with severe depression, bipolar disorder, pregnant,
* Subjects who are pregnant, attempting to get pregnant, or breast feeding
* Subjects with a known allergy or sensitivity to any component of the study ingredients.
* Subjects that do not understand the purpose and aspects of the study, do not sign the consent and do not complete the required treatment and follow up visit will also be excluded.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Self- perception of mood before treatment and after achieving an optimal cosmetic result as determined by the PI. | 1 month
  Treatment with Botox into the glabellar furrows increase the self- satisfaction with appearance once optimal correction is achieved beyond baseline in non -naïve users as compared to a control group and to themselves.
Happiness levels before treatment and after achieving an optimal cosmetic result as determined by the PI. | 1 month
  Treatment with Botox into the glabellar furrows increase the happiness levels once optimal correction is achieved beyond baseline in non -naïve users as compared to a control group and to themselves.

SECONDARY OUTCOMES:
Measurement of the Glabellar Wrinkle Severity Scores before treatment. The onset of effect and maximum efficacy compared to previous BOTOX Cosmetic injections will also be assessed by questionnaires. | 1 month
  Do non-naïve patients of Botox who have a baseline wrinkle severity score of 2 or 3 on the severity scale following an extended interval since last treatment of greater than 20 weeks achieve a two-point improvement 2 to 4 weeks after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dayan SH. Mind, Mood, and Aesthetics. Aesthet Surg J. 2015 Aug;35(6):759-61. doi: 10.1093/asj/sjv032. Epub 2015 Jun 4. No abstract available. PMID 26044342